CLINICAL TRIAL: NCT00955019
Title: Novel Method of Surveillance in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Kenneth K. Wang, M.D., Mayo Clinic
Other Study IDs: 07-002322; CA122426; NCT00629109 (obsolete NCT alias)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Barrett Esophagus
Keywords: Barrett's; Esophagus; Reflux; dysplasia; adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cytology specimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is being done to see how biomarkers (abnormalities in molecules of cells ) present in their Barrett's esophagus agree with results from surveillance biopsies; and to compare three different brush devices used to collect cells to see which of these 3 brush devices obtains a higher number of cells.

DETAILED DESCRIPTION:
During an endoscopy done for clinical surveillance of your Barrett's Esophagus participants are randomized to one of three brush devices by random chance like a flip of a coin. This is being done to see if one collects more cells than the others. A soft brush will be used to collect cells from the lining of the esophagus, this is known as brush cytology. With the endoscope positioned in your esophagus, samples (biopsies) of lining of the esophagus will then be taken to determine the nature of the Barrett's mucosa in the same manner as for any patient undergoing routine surveillance endoscopy for Barrett's esophagus. A part of the specimen will be used to store tissue samples that can later be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient age greater than 18 years of age
* Prior histological demonstration of Barretts Esophagus that is endoscopically visible with no dysplasia
* Low grade, high grade dysplasia or early esophageal cancer

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with barretts esophagus
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States